CLINICAL TRIAL: NCT05564741
Title: Hemodynamic Effects During Fast vs Slow Injection Time of Spinal Anaesthesia in Elderly Patients With Acute Hip Fracture .
Brief Title: Acute Hip Fracture and Spinal Anaesthesia Injection Time
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bengt Nellgard, Professor, Head of department, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Spinal time
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Hypotension; Hip Fractures; Anesthesia
Keywords: hip fracture; spinal anesthesia; hypotension; injection time
MeSH Terms: conditions — Hypotension; Hip Fractures | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 15 s injection time (Active Comparator): Patients in group A will be given the spinal anesthesia with an injection time of 15 s
  Interventions: Drug: Norepinephrine 1 MG/ML
- 90 s injection time (Active Comparator): Patients in group B will be given the spinal anesthesia with an injection time of 90 s
  Interventions: Drug: Norepinephrine 1 MG/ML

INTERVENTIONS:
Drug: Norepinephrine 1 MG/ML — As proxy for hypotension we record amount of Norepinephrine given during the study time of 30 minutes

SUMMARY:
The systemic effects of spinal anesthesia is not fully known. Our aim of this study is to assess whether there is a difference in hemodynamic effects if the spinal dose is given fast (15s) or slow (90s) in elderly patients with acute hip fracture (AHF). Ninety (n=90) patients with AHF planned for surgery within 72h at our hospital will be enrolled in the study and randomly devided into two groups. The patients will receive one predetermined dose of spinal anesthesia followed by an advanced minimally-invasive hemodynamic monitoring through an arterial line using FloTrac-system. The hemodynamic parameters will be conducted 10 minutes prior to the spinal anaesthesia and 30 minutes after the spinal block is given. Hypotension was defined as a fall in MAP > 30 % or a MAP <65mmHg.

DETAILED DESCRIPTION:
Both general and spinal anesthesia is known for inducing hypotension, which may be a problem for the elderly patients, often with many co-morbidities, causing a risk of organ hypoperfusion. At our clinic the investigators have a great experience with the neuraxial technique when operating these patients. Based on clinical experience the investigators hypothesise that a slow injection rate of the spinal dos would reduce the incidence and degree of hypotension. The investigators also aim to study the changes in the hemodynamic response between the groups in more detail as mentioned below.

Patients planned for acute hip fracture surgery in spinal anaesthesia at our hospital and fulfills the inclusion criteria will be included in our study. The investigators plan to include 90 patients, randomized in two groups where Group A will be given a spinal anaesthesia in 15s and Group B in 90s.

After arriving to the preoperative area, the patients will be given 5 L oxygen on a face mask and a standard monitoring with ECG, pulse- oximetry will be started, followed by the placement of a venous cannula and a radial arterial line. The patients will also be given a fascia iliaca compartment block (FIC) with ropivacaine 3,75 mg/ml 35-40 ml for comfort. In addition, the FloTrac system will be set up, using the existing arterial line, for advanced hemodynamic monitoring including invasive mean arterial pressure (MAP), Cardiac Index (CI), Heart Rate (HR), Stroke Volume (SV) and System Vascular Resistance (SVR)/ (SVRI).

A lumbal spinal anesthesia will be performed using a 25G pencil point needle. The intrathecal dose of anesthesia consists of isobar bupivacaine 5mg/ml 2,4 ml and fentanyl 50ug/ml 0,4ml. Sensory level will be monitored by "cold spray" Hypotension will be defined as a fall in MAP by >30% or MAP < 65 mmHg. As an surrogate factor for the aggregated time of hypotension the total amount of given vasopressor will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. >65 years of age
2. patient with hip fracture
3. ASA >/=2
4. scheduled for acute surgery in spinal anesthesia, 5. mentally intact to give informed consent

Exclusion Criteria:

1. anticoagulantion medication
2. planned for general anesthesia
3. surgery delayed > 72h
4. lack of informed consent.
5. severe aortic stenosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Mean arterial pressure (MAP) | 10 minutes before and 45 minutes after the intrathecal dose is given
  change in MAP after spinal anesthesia

SECONDARY OUTCOMES:
Cardiac Output (CO) | 10 minutes before and 45 minutes after the intrathecal dose is given
  CO change over time and relation to the speed of injection of the spinal anesthesia
Systemic vascular resistance over time and relation to the speed of injection of the spinal anesthesia | 10 minutes before and 45 minutes after the intrathecal dose is given

CONTACTS AND LOCATIONS:
Overall Officials: Bengt MD Nellgård, Prof, Study Director — Sahlgrenska University Hospital /Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffiths R, Babu S, Dixon P, Freeman N, Hurford D, Kelleher E, Moppett I, Ray D, Sahota O, Shields M, White S. Guideline for the management of hip fractures 2020: Guideline by the Association of Anaesthetists. Anaesthesia. 2021 Feb;76(2):225-237. doi: 10.1111/anae.15291. Epub 2020 Dec 2. PMID 33289066
- [Background] Nakasuji M, Suh SH, Nomura M, Nakamura M, Imanaka N, Tanaka M, Nakasuji K. Hypotension from spinal anesthesia in patients aged greater than 80 years is due to a decrease in systemic vascular resistance. J Clin Anesth. 2012 May;24(3):201-6. doi: 10.1016/j.jclinane.2011.07.014. PMID 22537572
- [Background] Wiles MD, Moran CG, Sahota O, Moppett IK. Nottingham Hip Fracture Score as a predictor of one year mortality in patients undergoing surgical repair of fractured neck of femur. Br J Anaesth. 2011 Apr;106(4):501-4. doi: 10.1093/bja/aeq405. Epub 2011 Jan 28. PMID 21278153
- [Background] Pitkanen M, Rosenberg P, Silvanto M, Tuominen M. Haemodynamic changes during spinal anaesthesia with slow continuous infusion or single dose of plain bupivacaine. Acta Anaesthesiol Scand. 1992 Aug;36(6):526-9. doi: 10.1111/j.1399-6576.1992.tb03512.x. PMID 1514336